CLINICAL TRIAL: NCT02225184
Title: The Impact of Delta Opioid Receptor Gene (OPRD1) Variations on Treatment Outcome in African Americans
Brief Title: Impact of Delta Opioid Receptor Gene (OPRD1) Variations on Treatment Outcome in African Americans
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914167; 14-DA-N167
Record Dates: First submitted 2014-08-23; First posted 2014-08-26 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2018-12-31

CONDITIONS: Genetic Underpinning of Substance Abuse; Polymorphism-genetic; Drug Abuse/Dependence; Opiod-Related Disorders
Keywords: Opioid Dependence; OPRM1; Outcome; Treatment
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other

SUMMARY:
Background:

- Differences in peoples genes can make them respond to drugs in different ways. Methadone and buprenorphine are two drugs used to treat drug addiction. A study showed that African Americans with a certain genetic marker did better using one kind of drug treatment over the other. Researchers want to see if they can repeat these findings. They also want to study other things that affect how well people do in treatment.

Objective:

- To see if certain genetic markers and other facts about a person s life can predict how well they do in treatment for addiction to opioids and cocaine.

Eligibility:

- African American adults age 18 and over. They must be former or current participants in an Archway Treatment Clinic study. They must have been on a stable dose of either study drug for at least 12 weeks. They also must have given urine samples regularly for at least 10 weeks.

Design:

* Participants will come to the clinic for 1 visit lasting about 2 hours.
* Participants will give 1 teaspoon of blood for genetic testing. They will be asked if their sample can be used in future studies.
* If researchers cannot get enough blood, they will do a cheek swab. This will collect skin cells for genetic testing.
* Participants will fill out 3 questionnaires.
* Results of genetic testing and answers to questionnaires will be kept private.

DETAILED DESCRIPTION:
The NIDA Clinical Trials Network s (CTN) START Study was designed to look at the pharmacogenetics of treatment response. The CTN investigators found that an intronic SNP (rs678849) in the gene for the opioid delta-1 receptor (OPRD1) strongly predicted treatment response in African-Americans. Specifically, during treatment with methadone, African-Americans with one variant of the SNP (CC) were less likely to use illicit opioids compared to African-Americans with other variants of the SNP (CT or TT) (relative risk = 0.53, 95% CI 0.46-0.60, p = 0.001). During treatment with buprenorphine, the association was reversed: African-Americans with the CC variant were more likely to use illicit opioids, compared to those with the CT or TT variants (relative risk = 2.13, 95% CI 1.81-2.45, p = 0.012). This pattern of findings was unexpected, both in terms of racial specificity and differential drug associations. Replication in a new sample is crucial to determining whether it represents a real effect.

Study objectives include: (1) To independently replicate the pharmacogenetic NIDA CTN findings by comparing urine drug screen opioid results for rs678849 genotype groups among opioid-addicted African-American individuals, treated with either buprenorphine or methadone; (2) To determine whether any effect of rs678849 genotype varies by demographic, drug use, mental health, and psychosocial characteristics; (3) To determine whether any effect of rs678849 genotype extends to cocaine use, and (4) To examine haplotype blocks in OPRD1 that might help explain the association.

We will recruit a sample of n=135 (to obtain 130 completers; 65 methadone, 65 buprenorphine) current and former participants in Archway treatment studies in order to have power of 0.80 to detect a difference of 0.5 standard deviations between rs678849 genotypes. To be eligible, participants must have received a stable dose (no taper > 7 days in length) of buprenorphine or methadone for at least 12 weeks and had at least 10 weekly urine drug screens during that time. After informed consent, in an approximate 3-hour session, participants will undergo collection of blood or a buccal swab for DNA extraction and analysis (blood is preferred, but buccal extraction enables inclusion of participants with poor venous access) and will complete 3 questionnaires; the Addiction Severity Index, the Perceived Neighborhood Scale, and sections of the Diagnostic Instrument for Genetic Studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Current or former participation in an Archway methadone or buprenorphine treatment study;
  2. Age 18 or older;
  3. Meet DSM-IV criteria for opioid dependence;
  4. Self-identified as African American, with at least 3 African American grandparents by self-report;
  5. At least 12 weeks of continuous treatment with a stable dose (no taper >7 days in length) of either buprenorphine or methadone, in a treatment regimen in which the physician considers dose increases in response to withdrawal symptoms, craving, or evidence of illicit opioid use by urine screens;
  6. At least 10 weeks of urine results available for analysis in that 12-week period, with no more than 6 consecutive urine data points missing, a requirement that should limit non-compliance as a factor;
  7. Able to speak and read English sufficiently to provide informed consent;
  8. Former participants only: have consented to future contact .

EXCLUSION CRITERIA:

(1) Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-08-23; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
To independently replicate the pharmacogenetic findings of the NIDA CTN START substudy by comparing urine opioid results as a function of rs678849 genotype among opioid-addicted African-Americans treated with either buprenorphine or methadone. | 9/2014 to 5/2016

CONTACTS AND LOCATIONS:
Overall Officials: Karran A Phillips, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States